CLINICAL TRIAL: NCT01371344
Title: A Long-term, Open-label, Non-comparative Study to Evaluate the Safety and Efficacy of a Modigraf® Based Immunosuppression Regimen in Paediatric Solid Allograft Recipients
Brief Title: A Paediatric, Open, Follow up Study With Modigraf Examining Safety and Efficacy in de Novo Allograft Recipients
Acronym: PROGRESSION
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Trial will not complete until at least 2025 and evolution of immunosuppressant therapy has made it unlikely that patients will convert from Modigraf to Prograf.
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F506-CL-0404; 2009-012259-21 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Heart Transplantation; Kidney Transplantation; Liver Transplantation
Keywords: Liver Transplantation; Kidney Transplantation; Heart Transplantation; Pharmacokinetics
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A: Heart Transplant (Tacrolimus granules) (Experimental): In Part A of the study, participants who are heart transplant recipients receive tacrolimus granules-based immunosuppressive regimen twice daily for a maximum of 1 year or until commercial availability of tacrolimus granules in the participant's country.
  Interventions: Drug: Tacrolimus granules
- Part A: Liver Transplant (Tacrolimus granules) (Experimental): In Part A of the study, participants who are liver transplant recipients receive tacrolimus granules-based immunosuppressive regimen twice daily for a maximum of 1 year or until commercial availability of tacrolimus granules in the participant's country.
  Interventions: Drug: Tacrolimus granules
- Part A: Kidney Transplant (Tacrolimus granules) (Experimental): In Part A of the study, participants who are kidney transplant recipients receive tacrolimus granules-based immunosuppressive regimen twice daily for a maximum of 1 year or until commercial availability of tacrolimus granules in the participant's country.
  Interventions: Drug: Tacrolimus granules
- Part B: All Participants (Tacrolimus capsules) (Experimental): In Part B of the study, participants who are heart, kidney or liver transplant recipients and who are converted from tacrolimus granules-based immunosuppression regimen, receive tacrolimus capsules twice daily for 1 month and thereafter receive commercially available tacrolimus capsules.
  Interventions: Drug: Tacrolimus capsules

INTERVENTIONS:
Drug: Tacrolimus granules — oral
  Other Names: Modigraf
  Arms: Part A: Heart Transplant (Tacrolimus granules); Part A: Kidney Transplant (Tacrolimus granules); Part A: Liver Transplant (Tacrolimus granules)
Drug: Tacrolimus capsules — oral
  Other Names: Prograf
  Arms: Part B: All Participants (Tacrolimus capsules)

SUMMARY:
The purpose of this study, a follow up to study FG506-CL-0403, is to see how safe and effective Modigraf® is (Part A) and to see how safe and effective it is to change your child's medication from Modigraf® to Prograf® (Part B).

DETAILED DESCRIPTION:
To monitor the safety and efficacy of Modigraf® (tacrolimus granules) in stable paediatric allograft recipients (Part A) and to monitor dose changes and tacrolimus whole blood trough levels after conversion from a Modigraf based Immunosuppression regimen to a Prograf® based Immunosuppression regimen (Part B).

ELIGIBILITY:
Inclusion Criteria:

F506-CL-0404 Part A

* Subject was ≤12 years of age at enrolment into study F506-CL-0403
* Subject received at least one dose of Modigraf in the F506-CL-0403 study

F506-CL-0404 Part B

* Subject received at least one dose of Modigraf in the F506-CL-0403 study
* Subject participated in F506-CL-0404 Part A
* Subject has continuously been dosed with Twice daily (BID) Modigraf since the End of Study Visit for Part A (ESVA) from F506-CL-0404 Part A
* Subject is stable and has had no dose changes in the preceding 2 weeks

Exclusion Criteria:

F506-CL-0404 Part A

* As all subjects included in this study conform to the exclusion criteria in study F506-CL-0403, hence no specific exclusion criteria are relevant for this study

F506-CL-0404 Part B

* There are no specific exclusion criteria for this study

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2011-06-24 (Actual); Primary Completion 2017-04-02 (Actual); Study Completion 2017-04-02 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants with Acute Rejection Episodes | Up to 12 months
  Rejection episodes/acute rejections are indicated by clinical and/or laboratory signs, and are classified according to their rejection specific treatment: •Spontaneously Resolving Acute Rejection: not treated with new or increased corticosteroid medication, antibodies or any other medication and resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Sensitive Acute Rejection: treated with new or increased corticosteroid medication only and which has resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Resistant Acute Rejection: did not resolve following treatment with corticosteroids; - Resolved with further treatment: any acute rejection with an end date AND a treatment other than corticosteroid used; - Unresolved with further treatment: any acute rejection with no end date AND a treatment other than corticosteroid used; - Unresolved with no further treatment: any acute rejection with no end date AND ONLY corticosteroid treatment used.
Part A; Number of Participants with Biopsy-proven Acute Rejection Episodes (BPARs) | Up to 12 months
  BPAR episodes are defined as acute rejection episodes confirmed by biopsy, and are classified according to their rejection specific treatment: •Spontaneously Resolving Acute Rejection: not treated with new or increased corticosteroid medication, antibodies or any other medication and resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Sensitive Acute Rejection: treated with new or increased corticosteroid medication only and which has resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Resistant Acute Rejection: did not resolve following treatment with corticosteroids; - Resolved with further treatment: any acute rejection with an end date AND a treatment other than corticosteroid used; - Unresolved with further treatment: any acute rejection with no end date AND a treatment other than corticosteroid used; - Unresolved with no further treatment: any acute rejection with no end date AND ONLY corticosteroid treatment used.
Part A: Severity of BPARs | Up to 12 months
  The severity of BPARs is categorized with specific criteria by organ: For kidney transplant participants, according to Banff '97 Diagnostic categories for renal allograft biopsies - Banff '07 update (C4d deposition, Acute antibody-mediated rejection I, II, and III, Acute T cell mediated rejection IA, IB, IIA, IIB and III); for liver transplant participants, according to 1997 Banff Schema for Grading of Liver Allograft Rejection - Rejection Activity Index score (sum of grades: 1-mild, 2-moderate, 3-severe; range from 0-9); for heart, according to Standardized Nomenclature of the International Society of Heart and Lung Transplantation - Standardised Cardiac Biopsy Grading: Acute Cellular Rejection 2004 (mild, moderate, severe).
Part A: Patient Survival | Up to 12 months
  Patient survival is reported as the number of deaths that occurred during Part A of the study.
Part A: Graft Survival | Up to 12 months
  Graft survival is reported as the number of participants who experienced graft loss. Graft loss is defined as retransplantation or death or return to pretransplantation treatment modality for 6 weeks or longer. Additionally, kidney transplanted participants with ongoing dialysis at the end of study is counted as participants with graft loss.
Part A: Number of Participants with Adverse Events (AEs) | From first dose of study drug up to 30 days after last dose of study drug (up to 13 months)
  Safety is assessed by AEs, which includes abnormalities identified during a medical test (e.g. clinical laboratory tests, vital signs, etc.) if the abnormality induces clinical signs or symptoms, needs active intervention, interruption or discontinuation of study medication or is clinically significant. A serious AE (SAE) is an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, is life-threatening, requires or prolongs hospitalization or is considered medically important. A treatment emergent adverse event (TEAE) is defined as an AE observed after investigational drug administration.
Part A: Tacrolimus Mean Trough Levels | Day 1, months 1, 2, 3, 6, 9, 12 (prior to each study drug dosing)
Part A: Number of Dose Adjustments | Months 1, 2, 3, 6, 9, 12
  Study drug doses are adjusted based on clinical evidence of efficacy and occurrence of adverse events, and taking into consideration the recommended whole blood trough level range of 5-20 ng/ml.
Part B: Number of Participants with AEs | From first dose of study drug (tacrolimus capsules) up to 7 days after last dose (up to 38 days)
  Safety is assessed by AEs, which included abnormalities identified during a medical test (e.g. clinical laboratory tests, vital signs, etc.) if the abnormality induces clinical signs or symptoms, needs active intervention, interruption or discontinuation of study medication or is clinically significant. A SAE is an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, is life-threatening, requires or prolongs hospitalization or is considered medically important. A TEAE is defined as an AE observed after investigational drug administration.
Part B: Tacrolimus Trough Levels Prior to and After Conversion | Day -1 up to 1 month
  Values prior to conversion are the last trough level prior to first dose of study drug (tacrolimus capsules). Values after conversion are the first trough level after first dose of study drug (tacrolimus capsules).
Part B: Number of Dose Adjustments | From first dose of study drug up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Senior Study Manager, Study Director — Astellas Pharma Europe Ltd.
Locations (12):
- Site BE40 Clinique Univ. Saint Luc, Brussels, Belgium
- France (2):
  - Site FR60 Groupement Hospitalier EST, Bron
  - Site FR61 Hopital Robert Debre, Paris
- Germany (2):
  - Site DE31 Kliniken der Medizinischen Hoc, Hanover
  - Site DE30 Universitätsklin Heidelberg, Heidelberg
- Site PL50 Centrum Zdrowia Dziecka, Warsaw, Poland
- Spain (4):
  - Site ES22 H.U. Gregorio Maranon, Madrid
  - Site ES20 Hospital Universitario La Paz, Madrid
  - Site ES21 Hospital Universitario La Paz, Madrid
  - Site ES23 Hospital Universitario La Paz, Madrid
- United Kingdom (2):
  - Site GB14 Alder Hey Children Hospital, Liverpool
  - Site GB13 Cent. Manchester Uni. Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=240